CLINICAL TRIAL: NCT04241783
Title: University of Bojnord
Brief Title: Relationship of Mindfulness, Artistic Activities and Quality of Life
Status: Completed | Type: Observational
Sponsor: Malahat Amani (Other)
Responsible Party: Sponsor-Investigator, Malahat Amani, assistant professor, University of Bojnord
Organization: University of Bojnord (Other)
Other Study IDs: 131809
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive — correlation

SUMMARY:
Methods: This study has the descriptive-correlational method and the statistical population was all artistic females of Bojnord city in 2018. In this study, 200 women of carpet weavers were selected by cluster random sampling. Participants filled out researcher-made questionnaires on how to do artistic activities, mindfulness, and quality of life. Data were analyzed using the Pearson correlation coefficient and hierarchical regression (moderator).

ELIGIBILITY:
Inclusion Criteria:

* be female, having 21 -60 years old, to work in workshops of weaving carpet, be literacy

Exclusion Criteria:

* be male, having under 21, upper 60, no work in workshops of weaving carpet , having psychotic disorders, be illiteracy

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation
Study Population: The study population consisted of women working in workshops of carpet weaving in Bojnourd in 2018 that were selected by cluster sampling from 5 workshops.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
quality of life | 3 day
  quality of life was measured by The World Health Organization Quality of Life. the questionnaire has 26 items measuring physical, psychological, social and environmental health factors. the items are also assessed on a 5-point scale. the high score on this questionnaire indicates a good quality of life.
mindfulness | 3 day
  mindfulness was measured by 39-item self-report scale made by Bauer et al (2006). this scale has observation, conscious action, non-judgmental of inner experience, description, and non-reaction factors. The items were assessed on a 5-point Likert scale. the high score on this scale indicates good mindfulness.
artistic activities | 3 day
  The researcher of this study designed seven items to measure the amount of artistic activity during the day and the week. the means of artistic activity is carpet weaving. a participant who is weaving carpet every day, she has high level artistic activities.

CONTACTS AND LOCATIONS:
Locations (1):
- university of Bojnord, Bojnourd, North Khorasan, Iran